CLINICAL TRIAL: NCT04745442
Title: Pilot Study of Antithrombin as Prophylaxis of Acute Respiratory Distress Syndrome in Patients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANTITROMBINA
Record Dates: First submitted 2021-02-08; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Severe Acute Respiratory Syndrome; Distress Respiratory Syndrome
Keywords: Antithrombin; COVID-19; Distress Respiratory Syndrome
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Pulmonary Atelectasis | interventions — Antithrombins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best available treatment + Antithrombin (Experimental): The subject will be treated with Antithrombin (50 IU/Kg/12h) for 72 hours and the best available treatment for COVID-19.
  Interventions: Drug: Antithrombin + best available treatment
- Best available treatment (Active Comparator): The subject will be treated with the best available treatment for COVID-19.
  Interventions: Drug: Best available treatment

INTERVENTIONS:
Drug: Antithrombin + best available treatment — The subject will be treated with Antithrombin (50 IU/Kg/12h) for 72 hours and the best available treatment for COVID-19.
  Arms: Best available treatment + Antithrombin
Drug: Best available treatment — The subject will be treated with the best available treatment for COVID-19.
  Arms: Best available treatment

SUMMARY:
Pilot clinical trial, with a marketed drug -natural component of human plasma-, not approved for this indication, single-center, exploratory, open, randomized, controlled, to study the efficacy and safety of human Antithrombin in patients with confirmed COVID-19 disease and criteria high risk to develop SARS.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 and < 85 years
* COVID-19 diagnosis confirmed.
* Radiological image compatible with COVID-19
* Present any of the following clinical-functional criteria considered RISK:

  1. Respiratory distress: Tachypnea > 26 breaths / minute
  2. PaO2 / FiO2 oxygenation index # 300
  3. Alteration of one or more of the following parameters:

  c.i. DD> 1,000 µg / L c.ii. Ferritin> 800 ng / mL 4.c.iii. Lymphocytes <800 cells / µL 4.c.iv. PCR> 100 mg / L 4.c.v. LDH> 500 U / L c.vi. IL-6> 15 pg / mL
* Direct or delegated verbal informed consent

Exclusion Criteria:

* Signs of active bleeding
* Immunosuppression by cancer or transplant
* Intolerance or allergy to AT or its components
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Combined variable: mortality or worsening rate with need for non-invasive mechanical ventilation or with need for invasive mechanical ventilation | At day 31 after randomization or hospital discharge (whichever occurs first)
  Combined variable: mortality or worsening rate with need for non-invasive mechanical ventilation or with need for invasive mechanical ventilation

SECONDARY OUTCOMES:
Time to clinical improvement (decreased risk of developing SARS or death) | At day 31 after randomization or hospital discharge (whichever occurs first)
  Time (in days) to improvement in the National Early Warning (NEWS) Score 2. Defined as the time, in days, from the start of treatment a two-point improvement on this scale.
Evaluate the improvement of the oxygenation index - PaO2 / FiO2- at 24 and 48 hours. | At 24 and 48 hours.
  Evaluate the improvement of the oxygenation index - PaO2 / FiO2- at 24 and 48 hours.
Improvement of the analytical parameters: time (in days) until the tendency to normalization (decrease >= 20%) of DD, ferritin, LDH, PCR and IL-6; the criteria reached before will be used. | At day 31 after randomization or hospital discharge (whichever occurs first)
  Improvement of the analytical parameters: time (in days) until the tendency to normalization (decrease >= 20%) of DD, ferritin, LDH, PCR and IL-6; the criteria reached before will be used.
Time (in days) until improvement in oxygenation: - Time until the SpO2 / FiO2 ratio exceeds the worst SpO2 / FiO2 prior to AT treatment. | At day 31 after randomization or hospital discharge (whichever occurs first)
  Time until the absence of oxygen need to maintain a basal saturation >= 92%.
Time to radiological improvement in radiological report. | At day 31 after randomization or hospital discharge (whichever occurs first)
  Time to radiological improvement in radiological report.
Time (in days) of non-invasive mechanical ventilation. | At day 31 after randomization or hospital discharge (whichever occurs first)
  Time (in days) of non-invasive mechanical ventilation.
Time (in days) of invasive mechanical ventilation. | At day 31 after randomization or hospital discharge (whichever occurs first)
  Time (in days) of invasive mechanical ventilation.
Mortality rate in hospital and one month after pharmacological intervention. | One month after pharmacological intervention.
  Mortality rate in hospital and one month after pharmacological intervention.
Percentage of patients who suffer any adverse effect related to pharmacological intervention. | One month after pharmacological intervention.
  Percentage of patients who suffer any adverse effect related to pharmacological intervention.
Incidence of adverse events related to medication and its administration. | At day 31 after randomization or hospital discharge (whichever occurs first)
  Incidence of adverse events related to medication and its administration.
Incidence in the appearance of allergic type hypersensitivity | At day 31 after randomization or hospital discharge (whichever occurs first)
  Incidence in the appearance of Acne, Generalized urticaria, Chest tightness, Dyspnoea, Hypotension and/or Anaphylaxis.
Incidence of B19 parvovirus infection | At day 31 after randomization or hospital discharge (whichever occurs first)
  Incidence of B19 parvovirus infection
Bleeding | At day 31 after randomization or hospital discharge (whichever occurs first)
  Incidence of Bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Salvatierra, MD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The information will be provided after the results are published in a journal.
Access Criteria: Upon request to uicec@imibic.org